CLINICAL TRIAL: NCT01950364
Title: A Phase 1 Study to Estimate MMAE Metabolites in Human Plasma and Urine in Patients With Relapsed or Refractory Classical Hodgkin Lymphoma or Relapsed or Refractory Systemic Anaplastic Large Cell Lymphoma Receiving Brentuximab Vedotin
Brief Title: A Phase 1 Study in Patients With Relapsed or Refractory Hodgkin Lymphoma or Systemic Anaplastic Large Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C25005; 2013-000193-29 (EudraCT Number); U1111-1174-1958 (Registry Identifier: WHO)
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-03

CONDITIONS: Hodgkin Lymphoma; Anaplastic Large-cell Lymphoma
Keywords: Lymphoma; Hodgkin; Anaplastic Large-cell; Relapsed; Refractory; Antigens, CD30; Antibody-Drug Conjugate; Antibodies, Monoclonal; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Anaplastic; Monomethyl auristatin E; Drug Therapy; Immunotherapy; Hematologic Diseases
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Lymphoma; Recurrence; Lymphoma, Non-Hodgkin; Hematologic Diseases | interventions — Brentuximab Vedotin; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Brentuximab vedotin (Experimental): Brentuximab vedotin will be administered every 3 weeks at a dose of 1.8 mg/kg.
  Interventions: Drug: brentuximab vedotin
- Arm B: Brentuximab vedotin and rifampicin (Experimental): Brentuximab vedotin will be administered every 3 weeks at a dose of 1.8 mg/kg beginning on Cycle 1, Day 1; daily rifampicin (600 mg PO) will be administered during Cycles 0 through 3 only, beginning on Cycle 0, Day 1 (7 days before the Cycle 1, Day 1 dose of brentuximab vedotin) and continuing through Cycle 3, Day 21.
  Interventions: Drug: Brentuximab vedotin and rifampicin

INTERVENTIONS:
Drug: brentuximab vedotin — Brentuximab vedotin will be administered every 3 weeks at a dose of 1.8 mg/kg.
  Other Names: SGN-35
  Arms: Arm A: Brentuximab vedotin
Drug: Brentuximab vedotin and rifampicin — Brentuximab vedotin will be administered every 3 weeks at a dose of 1.8 mg/kg beginning on Cycle 1, Day 1; daily rifampicin (600 mg PO) will be administered during Cycles 0 through 3 only, beginning on Cycle 0, Day 1 (7 days before the Cycle 1, Day 1 dose of brentuximab vedotin) and continuing through Cycle 3, Day 21.
  Other Names: SGN-35
  Arms: Arm B: Brentuximab vedotin and rifampicin

SUMMARY:
This is an open-label trial to estimate the concentrations of brentuximab vedotin in relapsed/refractory Hodgkin lymphoma (HL) or relapsed/refractory systemic anaplastic large cell lymphoma (sALCL) participants treated with either brentuximab vedotin or brentuximab vedotin + rifampicin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between 18 years and 75 years old, with relapsed or refractory HL or relapsed or refractory sALCL who have previously received at least 1 multiagent chemotherapy
* Measurable disease
* An Eastern Cooperative Oncology Group (ECOG) performance of 0 or 1
* Female participants who are postmenopausal for at least 1 year before the screening visit, surgically sterile, or agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 30 days after the last dose of study drug, or agree to practice true abstinence
* Male participants who agree to practice effective barrier contraception during the entire study treatment period through 6 months after the last dose of study drug or agree to practice true abstinence
* Clinical laboratory values as specified in the study protocol

Exclusion Criteria:

* Participants for whom rifampicin is contraindicated
* Previously received an allogeneic transplant.
* Participants with current diagnosis of primary cutaneous anaplastic large cell lymphoma (ALCL) (participants whose ALCL has transformed to sALCL are eligible).
* Known cerebral/meningeal disease including signs or symptoms of progressive multifocal leukoencephalopathy (PML)
* Female participants who are lactating and breastfeeding or pregnant
* Known human immunodeficiency virus (HIV) positive,
* Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (6):
- Belgium (2):
  - Brussels
  - Ghent
- Vilnius, Lithuania
- Spain (3):
  - Barcelona
  - Madrid
  - Salamanca

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in Belgium, Lithuania and Spain from 27 November 2013 to 16 June 2015.
Pre-assignment Details: Participants with a historical diagnosis of relapsed or refractory classical hodgkin lymphoma (HL) or relapsed or refractory systemic anaplastic large cell lymphoma (sALCL) were enrolled in 1 of 2 treatment groups: Brentuximab vedotin; Brentuximab vedotin + Rifampicin.
Groups:
- Brentuximab Vedotin: Brentuximab vedotin 1.8 milligram per kilogram (mg/kg), injection, intravenously, every 3 weeks on Day 1 of each 21-day treatment cycle up to a maximum of 16 brentuximab vedotin doses.
- Brentuximab Vedotin + Rifampicin: Brentuximab vedotin 1.8 mg/kg, injection, intravenously, every 3 weeks on Day 1 of each 21-day treatment cycle up to a maximum of 16 brentuximab vedotin doses and rifampicin, 600 milligram (mg), capsules, orally, once daily from Day 1 of treatment Cycle 0 through Day 21 of treatment cycle 3.
Period: Overall Study
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Started | 10 | 10
Completed | 0 | 0
Not Completed | 10 | 10
Not completed — Adverse Event | 3 | 0
Not completed — Stem Cell Transplant | 2 | 6
Not completed — Disease Progression | 5 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study drug.
Groups:
- Brentuximab Vedotin: Brentuximab vedotin 1.8 mg/kg, injection, intravenously, every 3 weeks on Day 1 of each 21-day treatment cycle up to a maximum of 16 brentuximab vedotin doses.
- Brentuximab Vedotin + Rifampicin: Brentuximab vedotin 1.8 mg/kg, injection, intravenously, every 3 weeks on Day 1 of each 21-day treatment cycle up to a maximum of 16 brentuximab vedotin doses and rifampicin, 600 mg, capsules, orally, once daily from Day 1 of treatment Cycle 0 through Day 21 of treatment cycle 3.
- Total: Total of all reporting groups
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (12.15) | 40.1 (9.13) | 41.2 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 7 | 4 | 11
Race/Ethnicity, Customized [Number; unit: participants]
  White | 10 | 10 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  Spain | 4 | 5 | 9
  Belgium | 2 | 1 | 3
  Lithuania | 4 | 4 | 8
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 71.11 (17.056) | 76.84 (24.213) | 73.98 (20.595)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 169.9 (3.80) | 169.7 (6.45) | 169.8 (5.15)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG performance status is used to assess how the disease affects the daily living abilities of the participant. It ranges on the scale from 0-5 (0= normal activity; 1= symptoms but ambulatory; 2= in bed for less than (<) 50 percent (%) of the time; 3= in bed for greater than (>) 50% of the time; 4= 100% bedridden; 5= dead.
  participants
    0 | 3 | 6 | 9
    1 | 6 | 4 | 10
    2 | 1 | 0 | 1
Disease Type [Number; unit: participants]
  Hodgkin lymphoma | 10 | 10 | 20
  sALCL | 0 | 0 | 0
Months from Initial Diagnosis to First Dose [Mean (Standard Deviation); unit: months] | 34.7 (31.23) | 61.9 (46.96) | 48.3 (41.25)
Ann Arbor Stage [Number; unit: participants] — Ann Arbor staging is staging system for lymphomas. The stage is determined by location of tumor. Stage I (located in a single region, usually 1 lymph node and surrounding area), Stage II (located in 2 separate regions, an affected lymph node or organ and a second affected area, and both affected areas are confined to 1 side of diaphragm), Stage III (spread to both sides of diaphragm, including organ/area near lymph nodes/spleen), Stage IV (diffuse or disseminated involvement of 1 or more extra lymphatic organs, including any involvement of liver, bone marrow or nodular involvement of lungs).
  participants
    I | 1 | 0 | 1
    II | 2 | 6 | 8
    III | 1 | 0 | 1
    IV | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 1, Predose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The lower limit of Quantification (LLQ) for all the observations was 0.01 nanogram/milliliter (ng/mL).
Time Frame: Cycle 1: Predose
Population: Pharmacokinetic (PK) analysis set included all participants who received brentuximab vedotin at 1.8 mg/kg throughout Cycles 1 to 3 and had sufficient dosing and PK data to reliably estimate PK parameters.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C4 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

2. Secondary Outcome: Serum Concentrations of Antibody-drug Conjugate (ADC)
Description: The LLQ for all the observations was 12.5 ng/mL.
Time Frame: Cycle 1 and 3: Predose, 0.5, 4, 72, 336 hours post-dose; Cycle 2: Predose, 0.5 hours post-dose; Cycle 3: 480 hours post-dose
Population: PK analysis set included all participants who received brentuximab vedotin at 1.8 mg/kg throughout Cycles 1 to 3 and had sufficient dosing and PK data to reliably estimate PK parameters.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  Cycle 1, Predose | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  Cycle 1, 0.5 hour | 29609.7759 (11865.35702) | 33125.0025 (10398.79403)
  Cycle 1, 4 hour | 24398.6482 (8092.41448) | 24533.2372 (6767.70744)
  Cycle 1, 72 hour | 4265.7542 (2880.39660) | 5958.0569 (1788.56378)
  Cycle 1, 336 hour | 1167.0713 (740.05650) | 1108.6515 (376.81123)
  Cycle 2, Predose | 794.3851 (10732.46886) | 435.1550 (303.25245)
  Cycle 2, 0.5 hour | 16032.6494 (15714.59821) | 31627.2566 (6716.71906)
  Cycle 3, Predose | 611.0573 (786.52082) | 536.3692 (524.72923)
  Cycle 3, 0.5 hour | 20991.9618 (12662.05087) | 33040.2245 (6295.45517)
  Cycle 3, 4 hour | 15378.8274 (9550.99903) | 24496.7203 (4212.84997)
  Cycle 3, 72 hour | 3258.7237 (3358.78504) | 4262.0364 (2431.24647)
  Cycle 3, 336 hour | 1381.2290 (1224.66857) | 1363.9488 (789.04877)
  Cycle 3, 480 hour | 648.2492 (1065.26404) | 734.5557 (634.23889)

3. Secondary Outcome: Serum Concentration of Total Antibody (TAb)
Description: The LLQ for all the observations was 12.5 ng/mL.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  Cycle 1, Predose | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  Cycle 1, 0.5 hour | 30874.4957 (11904.18494) | 30884.9074 (9956.67036)
  Cycle 1, 4 hour | 28577.3869 (9365.88746) | 28865.4674 (8192.50406)
  Cycle 1, 72 hour | 9931.2943 (4973.74692) | 11626.2147 (4396.55604)
  Cycle 1, 336 hour | 2898.2924 (1831.73997) | 3066.5859 (1017.84204)
  Cycle 2, Predose | 2055.3871 (10312.91280) | 1363.8319 (904.27346)
  Cycle 2, 0.5 hour | 17378.2105 (17543.51968) | 31583.7793 (7742.69918)
  Cycle 3, Predose | 1361.3147 (1592.89993) | 1517.6506 (1200.68646)
  Cycle 3, 0.5 hour | 15974.3723 (12467.10368) | 33892.4731 (10595.70675)
  Cycle 3, 4 hour | 11609.1430 (14719.69968) | 27548.1773 (7219.71925)
  Cycle 3, 72 hour | 13594.2016 (7492.70742) | 9588.9374 (5665.38218)
  Cycle 3, 336 hour | 3206.6925 (3000.22116) | 3628.9175 (1802.66091)
  Cycle 3, 480 hour | 1329.0886 (2024.17213) | 1866.5746 (1326.12113)

4. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 2, Predose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 2: Predose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 0.0919 (0.05695) | 0.0795 (0.14220)
  C4 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

5. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 3, Predose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 3: Predose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 0.1046 (0.10840) | 0.0727 (0.05936)
  C4 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

6. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 1, 0.5 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 1: 0.5 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 0.3902 (1.33635) | 0.2149 (0.43900)
  C4 | 0.0184 (0.00613) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0267 (0.02119) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C13 | 0.0108 (0.00360) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

7. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 2, 0.5 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 2: 0.5 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 0.3119 (1.69249) | 0.2929 (1.39185)
  C4 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | 0.0228 (0.00760)
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

8. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 3, 0.5 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 3: 0.5 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 0.3307 (2.33539) | 0.2577 (0.26736)
  C4 | 0.0256 (0.00905) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0323 (0.03266) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C13 | 0.0210 (0.00742) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

9. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 1, 4 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 1: 4 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 2.2778 (4.42089) | 1.7836 (0.93129)
  C4 | 0.0547 (0.02737) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | 0.0254 (0.01326) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | 0.0195 (0.01293) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0557 (0.05631) | 0.0160 (0.00921)
  C13 | 0.0151 (0.00752) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

10. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 3, 4 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 3: 4 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 1.7171 (4.42914) | 1.4529 (1.36620)
  C4 | 0.0397 (0.01323) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | 0.0163 (0.00804) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | 0.0118 (0.00600) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0446 (0.05011) | 0.0190 (0.01265)
  C13 | 0.0191 (0.00637) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

11. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 1, 24 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 1: 24 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 3.7950 (4.12446) | 3.1227 (2.38909)
  C4 | 0.0443 (0.05328) | 0.0191 (0.00637)
  C5 | 0.0218 (0.02814) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | 0.0206 (0.01477) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0805 (0.06986) | 0.0196 (0.01702)
  C13 | 0.0142 (0.00660) | 0.0113 (0.00377)

12. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 3, 24 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 3: 24 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 3.2336 (2.26369) | 2.2558 (1.60345)
  C4 | 0.0200 (0.01071) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | 0.0203 (0.01109) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | 0.0164 (0.00868) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0715 (0.04523) | 0.0177 (0.01284)
  C13 | 0.0105 (0.00371) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

13. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 1, 48 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 1: 48 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 4.2140 (3.69470) | 3.3727 (2.61792)
  C4 | 0.0424 (0.05259) | 0.0128 (0.00565)
  C5 | 0.0168 (0.02553) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | 0.0187 (0.01608) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0959 (0.06780) | 0.0210 (0.01455)
  C13 | 0.0134 (0.00763) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

14. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 3, 48 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 3: 48 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 3.4733 (2.17792) | 2.2156 (1.70890)
  C4 | 0.0193 (0.01407) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | 0.0198 (0.01316) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | 0.0170 (0.01112) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0746 (0.06162) | 0.0195 (0.01114)
  C13 | 0.0124 (0.00438) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

15. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 1, 72 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 1: 72 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 3.8931 (3.61834) | 3.0948 (2.03516)
  C4 | 0.0501 (0.06242) | 0.0127 (0.00423)
  C5 | 0.0190 (0.02664) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | 0.0241 (0.01640) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0899 (0.06688) | 0.0187 (0.01111)
  C13 | 0.0133 (0.00644) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

16. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 3, 72 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 3: 72 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 3.3047 (2.14127) | 1.9732 (1.32391)
  C4 | 0.0310 (0.01563) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | 0.0256 (0.01510) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | 0.0168 (0.01126) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0728 (0.04348) | 0.0187 (0.01079)
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

17. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 1, 96 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 1: 96 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 2.9148 (1.70500) | 3.2956 (2.97022)
  C4 | 0.0136 (0.00481) | 0.1420 (0.04733)
  C5 | 0.0120 (0.00643) | 0.0593 (0.01977)
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | 0.0374 (0.01247)
  C8 | 0.0660 (0.04349) | 0.0228 (0.06198)
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | 0.0108 (0.00360)

18. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 3, 96 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 3: 96 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 2.4449 (1.44334) | 2.2344 (1.81211)
  C4 | 0.0140 (0.00704) | 0.0418 (0.01393)
  C5 | 0.0205 (0.01017) | 0.0294 (0.00980)
  C7 | 0.0121 (0.00428) | 0.0252 (0.00840)
  C8 | 0.0622 (0.04328) | 0.0392 (0.04163)
  C13 | 0.0105 (0.00371) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

19. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 1, 144 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 1: 144 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 2.3326 (1.45619) | 1.7990 (0.89695)
  C4 | 0.0297 (0.02569) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | 0.0174 (0.01006) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | 0.0196 (0.00693) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0497 (0.02722) | 0.0120 (0.00542)
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

20. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 3, 144 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 3: 144 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 2.0555 (1.07315) | 1.2920 (0.75690)
  C4 | 0.0198 (0.00976) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | 0.0140 (0.00760) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | 0.0137 (0.00484) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0441 (0.02147) | 0.0145 (0.00648)
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

21. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 1, 336 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 1: 336 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 0.3130 (0.15743) | 0.2723 (0.16544)
  C4 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0127 (0.00672) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

22. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 3, 336 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 3: 336 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 0.4258 (0.30565) | 0.2578 (0.10847)
  C4 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0168 (0.01011) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

23. Primary Outcome: Plasma Concentration of Monomethylauristatin E (MMAE) and Its Metabolites at Cycle 3, 480 Hour Postdose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. The LLQ for all the observations was 0.01 ng/mL.
Time Frame: Cycle 3: 480 hour postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng/mL
  MMAE | 0.1189 (0.15808) | 0.0941 (0.03974)
  C4 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0114 (0.00431) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

24. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly; or a medically important event. AEs included both SAE and non-SAE.
Time Frame: Baseline up to 30 days after last dose of study drug (30 days after Cycle 16)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 10 | 10
participants
  AEs | 9 | 9
  SAEs | 4 | 0

25. Secondary Outcome: Number of Participants With Anti-therapeutic Antibodies (ATA) to Brentuximab Vedotin
Description: Participants with positive ATA at both Cycle 1 and 3, negative ATA at both Cycle 1 and 3, and transient positive (positive at one time point, but negative at the other) ATA for brentuximab vedotin were reported.
Time Frame: Day 1 of Cycle 1 and 3
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 10 | 10
participants
  Negative in both Cycle 1 and 3 | 5 | 7
  Positive in both Cycle 1 and 3 | 1 | 0
  Transient Positive | 2 | 2

26. Secondary Outcome: Number of Participants With Markedly Abnormal Laboratory Values
Description: The number of participants with any markedly abnormal standard safety laboratory values collected throughout study.
Time Frame: Baseline up to 30 days after last dose of study drug (30 Days after Cycle 16)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 10 | 10
participants | 5 | 5

27. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 1, Predose
Description: Metabolites of MMAE includes C4, C5, C7, C8 and C13. Amount of MMAE and its metabolites in urine were determined by multiplying the volume of urine obtained and the concentration of MMAE and its metabolites present in it, respectively. The LLQ for determining the concentration was 0.01 ng/mL.
Time Frame: Cycle 1: Predose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | 7.8900 (2.63000)
  C4 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | 0.0712 (0.02373)
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

28. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 1, 0-24 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 1: 0-24 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 12.5668 (5.31374) | 12.5020 (6.85958)
  C4 | 0.0878 (0.13223) | 0.0521 (0.02335)
  C5 | 0.0883 (0.10135) | 0.0254 (0.00847)
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.5967 (0.56221) | 0.1047 (0.07785)
  C13 | 0.0786 (0.11460) | 0.0456 (0.03714)

29. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 1, 24-48 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 1: 24-48 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 12.6225 (6.93735) | 11.7995 (6.20286)
  C4 | 0.0690 (0.10935) | 0.0392 (0.03010)
  C5 | 0.0863 (0.09138) | 0.0277 (0.01700)
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.7275 (0.59716) | 0.1568 (0.08381)
  C13 | 0.0722 (0.07482) | 0.0405 (0.03473)

30. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 1, 48-72 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 1: 48-72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 12.4089 (4.49922) | 11.6600 (5.45329)
  C4 | 0.0812 (0.15006) | 0.0419 (0.02694)
  C5 | 0.0867 (0.10841) | 0.0322 (0.01859)
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.7973 (0.38226) | 0.1189 (0.08494)
  C13 | 0.0786 (0.05672) | 0.0382 (0.02718)

31. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 1, 72-96 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 1: 72-96 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 10.7766 (8.14858) | 12.8426 (5.93538)
  C4 | 0.0867 (0.16449) | 0.0427 (0.02848)
  C5 | 0.0882 (0.11202) | 0.0394 (0.02131)
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.7480 (0.61219) | 0.1247 (0.08379)
  C13 | 0.0754 (0.06820) | 0.0415 (0.02723)

32. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 1, 96-120 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 1: 96-120 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 10.8018 (12.03431) | 9.5626 (7.26020)
  C4 | 0.0885 (0.11811) | 0.0414 (0.03529)
  C5 | 0.1053 (0.10639) | 0.0406 (0.02753)
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.7360 (1.02417) | 0.1034 (0.10563)
  C13 | 0.0630 (0.08155) | 0.0380 (0.03436)

33. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 1, 120-144 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 1: 120-144 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 6.7161 (6.13997) | 7.9830 (4.33309)
  C4 | 0.0730 (0.08387) | 0.0335 (0.02037)
  C5 | 0.0836 (0.07377) | 0.0301 (0.01767)
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.4477 (0.56047) | 0.0910 (0.06044)
  C13 | 0.0551 (0.05107) | 0.0345 (0.01738)

34. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 1, 144-168 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 1: 144-168 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 5.5693 (3.50945) | 5.8025 (3.45889)
  C4 | 0.0579 (0.06807) | 0.0448 (0.02158)
  C5 | 0.0747 (0.05078) | 0.0287 (0.01527)
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.3916 (0.34491) | 0.0706 (0.03027)
  C13 | 0.0438 (0.03146) | 0.0363 (0.01283)

35. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 1, 336-360 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 1: 336-360 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 1.0727 (0.55233) | 1.3326 (0.80959)
  C4 | 0.0459 (0.01530) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | 0.0289 (0.00963) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0751 (0.04505) | 0.0401 (0.02242)
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

36. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 1, 480-504 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 1: 480-504 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 0.4420 (0.30745) | 0.3505 (0.14592)
  C4 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0578 (0.03314) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

37. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 3, Predose
Description: as for outcome 27
Time Frame: Cycle 3: Predose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 0.3171 (0.33548) | 0.4227 (0.17918)
  C4 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0392 (0.02985) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

38. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 3, 0-24 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 3: 0-24 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 10.7174 (15.35912) | 12.4438 (8.86144)
  C4 | 0.0454 (0.07644) | 0.0451 (0.02977)
  C5 | 0.0509 (0.04623) | 0.0301 (0.01847)
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.4657 (0.41352) | 0.1285 (0.17930)
  C13 | 0.0516 (0.07045) | 0.0676 (0.05022)

39. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 3, 24-48 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 3: 24-48 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 11.1360 (6.73693) | 13.2483 (4.79482)
  C4 | 0.0604 (0.05049) | 0.0413 (0.03095)
  C5 | 0.0808 (0.06838) | 0.0311 (0.02021)
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.5750 (0.58196) | 0.1600 (0.11946)
  C13 | 0.0637 (0.05102) | 0.0507 (0.03607)

40. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 3, 48-72 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 3: 48-72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 12.7267 (8.96991) | 13.8072 (8.63973)
  C4 | 0.0620 (0.06222) | 0.0524 (0.04691)
  C5 | 0.0746 (0.09237) | 0.0406 (0.03034)
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.6950 (0.83588) | 0.1598 (0.14846)
  C13 | 0.0632 (0.06480) | 0.0746 (0.05134)

41. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 3, 72-96 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 3: 72-96 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 11.2527 (8.65574) | 12.2263 (6.09003)
  C4 | 0.0702 (0.07079) | 0.0611 (0.05055)
  C5 | 0.0937 (0.10757) | 0.0437 (0.03084)
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.5276 (0.95507) | 0.1510 (0.11532)
  C13 | 0.0573 (0.07734) | 0.0564 (0.03759)

42. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 3, 96-120 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 3: 96-120 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 8.3817 (7.78279) | 8.1426 (7.29530)
  C4 | 0.0710 (0.05912) | 0.0512 (0.04137)
  C5 | 0.0916 (0.08893) | 0.0435 (0.02885)
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.5198 (0.79634) | 0.1088 (0.09569)
  C13 | 0.0607 (0.06838) | 0.0524 (0.03619)

43. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 3, 120-144 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 3: 120-144 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 7.3500 (3.78427) | 7.5871 (4.66863)
  C4 | 0.0461 (0.03666) | 0.0520 (0.03870)
  C5 | 0.0657 (0.04811) | 0.0342 (0.02508)
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.4700 (0.37131) | 0.0869 (0.07672)
  C13 | 0.0386 (0.03212) | 0.0429 (0.02820)

44. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 3, 144-168 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 3: 144-168 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 6.1125 (3.83207) | 4.6823 (2.80767)
  C4 | 0.0538 (0.04252) | 0.0562 (0.02674)
  C5 | 0.0662 (0.06110) | 0.0308 (0.01718)
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.3485 (0.45898) | 0.0651 (0.03984)
  C13 | 0.0402 (0.04117) | 0.0481 (0.01603)

45. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 3, 336-360 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 3: 336-360 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 1.2811 (1.55068) | 0.8271 (0.43597)
  C4 | 0.0377 (0.01812) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | 0.0347 (0.02457) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0734 (0.10958) | 0.0277 (0.01306)
  C13 | 0.0227 (0.00757) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

46. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included body temperature, body weight, blood pressure and heart rate.
Time Frame: Baseline up to 30 days after last dose of study drug (30 Days after Cycle 16)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 10 | 10
participants | 1 | 2

47. Primary Outcome: Amount of Monomethylauristatin E (MMAE) and Its Metabolites Excreted in Urine at Cycle 3, 480-504 Hours Postdose
Description: as for outcome 27
Time Frame: Cycle 3: 480-504 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Number analyzed (Participants) | 9 | 9
ng
  MMAE | 0.4660 (0.41713) | 0.3334 (0.25074)
  C4 | 0.0248 (0.00827) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C5 | 0.0377 (0.01257) | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C7 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.
  C8 | 0.0620 (0.04967) | 0.0221 (0.00737)
  C13 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported. | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol results were to be summarized only for observations above LLQ, hence, data was not reported.

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (30 days after Cycle 16).
Description: Serious and non-serious AEs were collected from first dose through 30 days after the last dose (Cycle 16). Beginning on Cycle 4 Day 1, only AEs with Grade 3 were recorded. Exceptions: New onset AEs of Grade 1-2 were recorded if they met criteria for SAEs or resulted in dose modification; PN events will be recorded regardless of severity grade.
Arm/Group | Brentuximab Vedotin | Brentuximab Vedotin + Rifampicin
Serious Adverse Events (participants affected / at risk) | 4/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin (N=10) | Brentuximab Vedotin + Rifampicin (N=10)
Thrombosis in device (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin (N=10) | Brentuximab Vedotin + Rifampicin (N=10)
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 3 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Eosinophilia (Blood and lymphatic system disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2
Pyrexia (General disorders) | 1 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 2
Fatigue (General disorders) | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Local swelling (General disorders) | 1 | 0
Localised oedema (General disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.